CLINICAL TRIAL: NCT04188548
Title: EMBER: A Phase 1a/1b Study of LY3484356 Administered as Monotherapy and in Combination With Anticancer Therapies for Patients With ER+ Locally Advanced or Metastatic Breast Cancer and Other Select Non-Breast Cancers
Brief Title: A Study of LY3484356 in Participants With Advanced or Metastatic Breast Cancer or Endometrial Cancer
Acronym: EMBER
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17502; J2J-MC-JZLA (Other: Eli Lilly and Company); 2019-003581-41 (EudraCT Number)
Record Dates: First submitted 2019-11-18; First posted 2019-12-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms | interventions — Imlunestrant; abemaciclib; Everolimus; Alpelisib; Trastuzumab; Aromatase Inhibitors; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation LY3484356 (Experimental): LY3484356 given orally.
  Interventions: Drug: LY3484356
- Part A: Dose Expansion: LY3484356 + Abemaciclib +/- AI (Experimental): LY3484356 and abemaciclib given orally in combination with or without Aromatase Inhibitor (AI) of physician's choice (Anastrozole, Exemestane, or Letrozole) administered orally.
  Interventions: Drug: LY3484356; Drug: Abemaciclib; Drug: Aromatase Inhibitor (AI)
- Part B: Dose Expansion: Cohort E3: LY3484356 (Experimental): LY3484356 given orally.
  Interventions: Drug: LY3484356
- Part B: Dose Expansion: Cohort E4: LY3484356 + Everolimus (Experimental): LY3484356 and everolimus given orally.
  Interventions: Drug: LY3484356; Drug: Everolimus
- Part B: Dose Expansion: Cohort E5: LY3484356 + Alpelisib (Experimental): LY3484356 and alpelisib given orally.
  Interventions: Drug: LY3484356; Drug: Alpelisib
- Part C:Dose Expansion: LY3484356 + Trastuzumab +/- Abemaciclib (Experimental): LY3484356 administered orally in combination with trastuzumab intravenously with or without Abemaciclib.
  Interventions: Drug: LY3484356; Drug: Abemaciclib; Drug: Trastuzumab
- Part D: Dose Expansion: LY3484356 +/- Abemaciclib (Experimental): LY3484356 and Abemaciclib given orally with trastuzumab administered intravenously.
  Interventions: Drug: LY3484356; Drug: Abemaciclib
- Part E: Dose Expansion: LY3484356 + Trastuzumab + Pertuzumab (Experimental): LY3484356 administered orally in combination with trastuzumab and pertuzumab administered intravenously.
  Interventions: Drug: LY3484356; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: LY3484356 — Administered orally
  Other Names: Imlunestrant
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Part A: Dose Expansion: LY3484356 + Abemaciclib +/- AI; Part C:Dose Expansion: LY3484356 + Trastuzumab +/- Abemaciclib; Part D: Dose Expansion: LY3484356 +/- Abemaciclib
Drug: Everolimus — Administered orally
  Arms: Part B: Dose Expansion: Cohort E4: LY3484356 + Everolimus
Drug: Alpelisib — Administered orally
  Arms: Part B: Dose Expansion: Cohort E5: LY3484356 + Alpelisib
Drug: Trastuzumab — Administered intravenously
  Arms: Part C:Dose Expansion: LY3484356 + Trastuzumab +/- Abemaciclib; Part E: Dose Expansion: LY3484356 + Trastuzumab + Pertuzumab
Drug: Aromatase Inhibitor (AI) — Anastrozole or Exemestane or Letrozole administered orally (physician choice)
  Arms: Part A: Dose Expansion: LY3484356 + Abemaciclib +/- AI
Drug: Pertuzumab — Administered intravenously
  Arms: Part E: Dose Expansion: LY3484356 + Trastuzumab + Pertuzumab

SUMMARY:
The reason for this study is to see if the study drug LY3484356 alone or in combination with other anticancer therapies is safe and effective in participants with advanced or metastatic breast cancer or endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

All study parts:

* Participants must be willing to provide adequate archival tissue sample
* Participants must be willing to use highly effective birth control
* Participants must have adequate organ function
* Participants must be able to swallow capsules

Dose escalation- Participants must have one of the following:

* Parts A and B: ER+ HER2- breast cancer with evidence of locally advanced unresectable or metastatic disease who have had the following:
* Part A: may have had up to 1 prior regimen of any kind for in the advanced/metastatic setting and no prior cyclin-dependent kinase 4/6 (CDK4/6) inhibitor therapy.
* Part B: may have had up to 2 prior regimens, no more than 1 of which may be endocrine therapy in the advanced/metastatic setting, and must have received a prior CDK4/6 inhibitor
* Cohort E4: No prior everolimus.
* Cohort E5: No prior alpelisib and must have a phosphatidylinositol 3-kinase catalytic α (PIK3Cα) mutation as determined by local testing.
* Part C: ER+, human epidermal growth factor receptor 2 positive (HER2+) breast cancer with evidence of locally advanced unresectable or metastatic disease who have had at least 2 HER2-directed therapies in any setting.
* Part D: ER+, EEC that has progressed after platinum containing chemotherapy and no prior fulvestrant or aromatase inhibitor therapy.
* Part E: ER+ and HER2+ breast cancer with evidence of locally advanced, unresectable, or metastatic disease.
* Part E: Participants must have received induction taxane chemotherapy combined with trastuzumab + pertuzumab as first-line treatment for advanced/metastatic disease and must not have progressed on this regimen.
* Part E: Participants must not have received more than 1 HER2-directed regimen or any endocrine therapy for advanced disease or any prior CDK4/6 inhibitor therapy.

Participants with ER+/HER2- breast cancer enrolled in this study must have had evidence of clinical benefit while on endocrine therapy for at least 24 months in the adjuvant setting or at least 6 months in the advanced/metastatic setting or have untreated de novo metastatic breast cancer

Exclusion Criteria:

* Participants must not have certain infections such as hepatitis or tuberculosis or HIV that are not well controlled
* Participants must not have another serious medical condition
* Participants must not have cancer of the central nervous system that is unstable
* Participants must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) and DLT-Equivalent Toxicities | Baseline through Cycle 1 (21/28 Day Cycle)
  Number of Participants with DLTs and DLT-Equivalent Toxicities

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3484356 | Predose Cycle 1 Day 1 through Predose Cycle 2 Day 1 (21/28 Day Cycles)
  PK: AUC of LY3484356
PK: Maximum Concentration (Cmax) of LY3484356 | Predose Cycle 1 Day 1 through Predose Cycle 2 Day 1 (21/28 Day Cycles)
  PK: Cmax of LY3484356
PK: AUC of LY3484356 in Combination with Other Anticancer Therapies | Predose Cycle 1 Day 1 through Predose Cycle 2 Day 1 (21/28 Day Cycles)
  PK: AUC of LY3484356 in Combination with Other Anticancer Therapies
PK: Cmax of LY3484356 in Combination with Other Anticancer Therapies | Predose Cycle 1 Day 1 through Predose Cycle 2 Day 1 (21/28 Day Cycles)
  PK: Cmax of LY3484356 in Combination with Other Anticancer Therapies
Overall Response Rate (ORR): Percentage of Participants with Confirmed Complete Response (CR) or Partial Response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline through Disease Progression or Death (Estimated up to 28 Months)
  ORR: Percentage of Participants with Confirmed CR or PR as per RECIST v1.1
Duration of Response (DoR): Time From the Date of First Evidence of CR, PR (per RESIST v1.1) to the Date of Objective Progression or Death Due to Any Cause, Whichever is Earlier | Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Estimated up to 28 Months)
  DoR: Time From the Date of First Evidence of CR, PR (per RESIST v1.1) to the Date of Objective Progression or Death Due to Any Cause, Whichever is Earlier
Disease Control Rate (DCR): Percentage of Participants with a Best Overall Response (BOR) of CR, PR, and Stable Disease (SD) as per RECIST v1.1 | Baseline through Measured Progressive Disease (Estimated up to 28 Months)
  DCR: Percentage of Participants with a BOR of CR, PR, and SD as per RECIST v1.1
Clinical Benefit Rate (CBR): Percentage of Participants with a BOR of CR or PR, or SD lasting ≥24 weeks as per RECIST v1.1 | Baseline through Measured Progressive Disease (Estimated up to 28 Months)
  CBR: Percentage of Participants with a BOR of CR or PR, or SD lasting ≥24 weeks as per RECIST v1.1
Progression Free Survival (PFS): Time From Baseline to the Date of Objective Progression or Death Due to Any Cause, Whichever is Earlier | Baseline to Objective Progression or Death Due to Any Cause (Estimated up to 28 Months)
  PFS: Time From Baseline to the Date of Objective Progression or Death Due to Any Cause, Whichever is Earlier

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (42):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of California, Irvine, Orange, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lake Nona DDU, Orlando, Florida
  - Winship Cancer Center Emory University, Atlanta, Georgia
  - Community Cancer Center North, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology/Hematology PA, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering - Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmot Cancer Institute, Rochester, New York
  - Duke University, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - UPMC Hillman Cancer Center Harrisburg, Harrisburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology Nashville, Nashville, Tennessee
  - UT Southwestern Med Center, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Minnesota Oncology/Hematology PA, The Woodlands, Texas
  - Oncology and Hematology Associates of Southwest Virginia Inc, The Woodlands, Texas
  - Texas Oncology - San Antonio Medical Center, The Woodlands, Texas
  - US Oncology, The Woodlands, Texas
  - USO-Rocky Mountain Cancer Center, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (5):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Breast Cancer Research Centre-WA, Nedlands, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
- Belgium (3):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Institut Jules Bordet, Anderlecht, Bruxelles-Capitale, Région de
  - UZ Leuven, Leuven, Vlaams-Brabant
- France (2):
  - Institut Curie, Paris
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
- Japan (2):
  - Hyogo Cancer Center, Akashi, Hyōgo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- South Korea (4):
  - Severance Hospital, Yonsei University Health System, Seoul, Korea
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clínico Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhave M, Jhaveri KL, Kaufman PA, Aftimos P, Lombard J, Giridhar KV, Im SA, Ma CX, Lee KT, Kim SB, Sohn J, Li Y, Yuen E, Estrem ST, Nguyen B, Makena MR, Ismail-Khan R, Beeram M. Imlunestrant, an oral selective estrogen receptor degrader, in combination with HER2 directed therapy, with or without abemaciclib, in ER-positive, HER2-positive advanced breast cancer: results from the phase 1a/1b EMBER study. Breast Cancer Res. 2025 Dec 21. doi: 10.1186/s13058-025-02168-6. Online ahead of print. No abstract available. PMID 41423595
- [Derived] Jhaveri KL, Lim E, Jeselsohn R, Ma CX, Hamilton EP, Osborne C, Bhave M, Kaufman PA, Beck JT, Manso Sanchez L, Parajuli R, Wang HC, Tao JJ, Im SA, Harnden K, Yonemori K, Dhakal A, Neven P, Aftimos P, Pierga JY, Lu YS, Larson T, Jerez Y, Sideras K, Sohn J, Kim SB, Saura C, Bardia A, Sammons SL, Bacchion F, Li Y, Yuen E, Estrem ST, Rodrik-Outmezguine V, Nguyen B, Ismail-Khan R, Smyth L, Beeram M. Imlunestrant, an Oral Selective Estrogen Receptor Degrader, as Monotherapy and in Combination With Targeted Therapy in Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Phase Ia/Ib EMBER Study. J Clin Oncol. 2024 Dec 10;42(35):4173-4186. doi: 10.1200/JCO.23.02733. Epub 2024 Sep 6. PMID 39241211
- See also: A Study of LY3484356 in Participants With Advanced or Metastatic Breast Cancer — https://trials.lillytrialguide.com/en-US/trial/2zSLrHO7ERDGXZvPbUVdZm